# CARISBAMATE AS A POTENTIAL TREATMENT FOR ALCOHOL DEPENDENCE

NCT02435381

ICF drafted June 13, 2017

The protocol was formally closed by the IRB on 9/18/2017



| Subject Name: | | Date: |
|---|---|---|
| Subject Initials: | | |
| Principal Investigator: | THOMAS F. NEWTON | VAMC: |
| H-30334 - CARISBAMATE | AS A POTENTIAL TREATMENT FOR AL | .COHOL DEPENDENCE |

#### standard consent

#### **Background**

You are invited to take part in a research study. Please read this information and feel free to ask any questions before you agree to take part in the study.

You are being asked to take part in this research study, carried out by the investigators listed at the end of this consent form because 1) you drink alcohol regularly and you are otherwise healthy; 2) you are 18-55 years of age; 3) you are not seeking treatment for alcohol use at this time.

Please read this information and feel free to ask any questions before you agree to take part in the study.

This study is a clinical research trial looking at the safety and effectiveness of a drug, called carisbamate, in combination with alcohol. Carisbamate is not approved by the FDA.

If you are seeking treatment, you should not participate in this study and the investigators can refer you to organizations that offer treatment for alcohol addiction.

This consent form has information that will be discussed with you about the purpose of this study, whether participation may benefit you, the risks of your participation, and what is expected of you. You should read the information below, and ask questions about anything you do not understand, before deciding whether or not to participate. Once you understand the study, and if you wish to participate, you will be asked to sign this consent form. You will be given a copy to keep. Your participation in this research study is totally VOLUNTARY, and you may decide not to participate, or decide to leave at any time. If you choose to not participate or drop out at any time, it will not affect your right to medical care at Baylor College of Medicine or Michael E. DeBakey Veterans Affairs Medical Center.

#### **Purpose**

The purpose of this study is to find out if carisbamate is a safe and effective medication to treat alcohol dependence.

#### **Procedures**

The research will be conducted at the following location(s): Baylor College of Medicine, Michael E. DeBakey Veterans Affairs Medical Center.

PRE-INTAKE SCREENING

The pre-intake screening described below may be scheduled over several visits within a 2-week period. Study procedures will last about 8 days, divided in two 4-day phases. All procedures will be done as an inpatient; you will be required to stay overnight in the hospital for 8 nights. Most participants

JAN 1990 10-1086

Last Amendment: 8/26/2013



| Subject Name: Subject Initials: | | Date: |
|---|---|---|
| Principal Investigator: | THOMAS F. NEWTON | VAMC: |
| H-30334 - CARISBAMAT | E AS A POTENTIAL TREATMENT FOR ALCOHOL DEF | PENDENCE |

spend their free time in the hospital reading, watching tv, and playing computer games.

Based on the results of the pre-intake screening, you may not be eligible to participate in the rest of this study.

If you are eligible and agree to participate in this study and sign this consent form, we will ask you to undergo the following research procedures:

During the pre-intake screening, you will answer a number of questions about your alcohol habit, history and present alcohol and use behavior, as well as about your mood and physical well-being. You will have your heart rate and blood pressure checked, and you will be asked questions concerning the type and quantity of prescribed and non-prescribed drugs you use. You have the right to refuse to answer any question that you may not wish to answer.

In order to determine if you are healthy enough to be in this study, you will have a physical exam and medical history taken by one of the study doctors. You will be asked for a 30cc (approximately 2 tablespoons) blood sample, to test that your liver

and kidneys are functioning normally and to test your blood to make sure it is normal and you do not have hepatitis.

You will have your heart checked with an electrocardiogram (ECG) at screening. The ECG will measure how your heart functions and check for heart problems or disease. For the ECG, a trained technician will attach a number of small electrodes (using a type of adhesive that is easily removed) to your body. Your heartbeats will then be recorded for about 1 minute, and the electrodes and adhesive will be removed. If signs of illness are detected, you will be told, referred to a list of physicians, and then excluded from the rest of the study.

You will also give a urine sample for drug testing. All urine samples will be destroyed after analysis. If you test positive for any illicit substances, you cannot participate in the study. You will take an alcohol breath test to see if there is any alcohol in your blood. You may still participate in the study if alcohol is present in your blood at the time of screening.

If more than 30 days go by after the screening visit before you are admitted to the study, the screening assessments will be repeated.

#### WOMEN OF CHILDBEARING POTENTIAL

If you are a woman of childbearing potential (being able to become pregnant), due to the possible risks to a fetus, you may not participate in this study unless you are not pregnant and, with the investigator's knowledge and approval, you are using a medically acceptable form of birth control (contraception). Examples of reliable forms of birth control include the Pill, Norplant, Depo-Provera, and consistent and

VA FORM **10-1086** JAN 1990



| Subject Name: | | Date: |
|---|---|---|
| Subject Initials: | | |
| Principal Investigator: | THOMAS F. NEWTON | VAMC: |
| H-30334 - CARISBAMATE | AS A POTENTIAL TREATMENT FOR ALCOHO | OL DEPENDENCE |

correct use of condoms. You must agree to give urine samples to test for pregnancy (at no charge to you) before entering the study, at each admission and when the study is over.

#### ADMISSION AND STUDY PROCEDURES

You will be admitted to the Research Commons unit at the Michael DeBakey VA medical center. For your safety, we request that you do not leave the research unit during the study. However, if a family emergency presents itself and you feel you must leave, the study doctor will consider these requests on a case-by-case basis.

For the duration of the study, you are required to stop drinking alcohol, apart from the study procedures. Upon admission to the hospital, your belongings will be searched for drugs and alcohol. While you are in the study, urine and breath alcohol level tests will be administered daily to ensure that you are compliant with the study rules. Visitors will not be allowed during your hospital stay. You will stay at the hospital for 8 days but scheduling and/or safety reasons may result in your staying a day or so extra.

On the first day of admission, you will complete a number of interviews and questionnaires on a computer, a few of which will be repeated daily to follow your progress. Interviews and questionnaires are used to measure your feelings, attitudes, and psychiatric and social history. Some will be given by the investigators, and some you will read and answer by yourself. The questionnaires and interviews on the day of admission will take up to 2 hours to complete. The daily questionnaires will take 10-15 minutes to complete.

## STUDY DRUGS

You will receive both carisbamate and placebo (an inactive pill like a sugar pill) during the study. You will not be told which pills you are taking on which days. On Day 1 you will start taking carisbamate 300mg or a sugar pill twice day. If you have any side effects (see below under Risk) syou must report them immediately to the study personnel, study doctor and

the floor nurses. A list of names is provided at the end of this document. You will take the last pills on day 4. Then you will have a week off. When you return to the clinic for phase 2 of the study, you will again take the study pills for 4 days.

#### Alcohol doses

On day 4 of each phase you will receive one beverage with alcohol and one without alcohol. During the procedures, you will sit and be relaxed and comfortable in a chair or bed. You will receive 0.8g/kg of alcohol which is a moderate dose, making most people feel "buzzed". Study staff will be present after you drink the alcohol to monitor your safety. You may not smoke cigarettes from 1-hour prior to session initiation until 90 minutes afterwards.

Your blood pressure and heart rate will be measured before, during, and after you drink the beverage

VA FORM JAN 1990 **1** 

10-1086

Last Amendment: 8/26/2013 BCM Approval from June 13, 2017 to June 12, 2018



| Subject Name: | | Date: |
|---|---|---|
| Subject Initials: | | |
| Principal Investigator: | THOMAS F. NEWTON | VAMC: |
| H-30334 - CARISBAMATI | E AS A POTENTIAL TREATMENT FOR AL | LCOHOL DEPENDENCE |

until they have returned to normal. Smoking will not be permitted within 15 minutes of scheduled vital sign measurements. Before and after drinking the alcohol, you will also be asked questions concerning your emotional and physical state, and to rate your alcohol craving. This will occur every half hour until 3 hours after you drink the beverages.

Before you are discharged from the study on day 4 of each phase, you will complete the end-of-study procedures, which include forms, and assessment to be medically stable by the study doctor. You can see and get a copy of your research related health information. However, your research doctor may be unable to provide you with a copy of your information until the end of the study.

## **Potential Risks and Discomforts**

You must tell the study doctor or nurse before enrolling in any other clinical trials while on this study.

## **RISKS OF STUDY DRUGS**

#### RISKS OF CARISBAMATE

Carisbamate has proven safe administered alone and in combination with other medications to treat seizure disorders. The most frequently reported side effect is dizziness. Other side effects may include sedation, headaches and changes in sensation.

#### **RISKS OF ALCOHOL**

Alcohol has a range of side-effects. Alcohol in small to moderate amounts can cause increased sociability, euphoria, drowsiness, and disorientation. Acute alcohol can compromise motor skills, impair judgment and alter cardiovascular measures.

#### RISKS OF CARISBAMATE AND ALCOHOL TOGETHER

It is possible that the risks of carisbamate and alcohol interact when they are given together; in other words, one could increase the effects of the other, although this is not expected.

#### RISKS OF BLOOD COLLECTION

The risks of inserting a needle into a vein may involve (1) pain from insertion of the needle; (2) lightheadedness; (3) fainting; (4) hematoma (like a bruise) at the site of the needle insertion; (5) inflammation of the vein; (6) clotting of the vein; (7) rarely, infection where the needle enters the skin, or (8) rarely, an allergic reaction to the tape applied afterwards.

## RISKS OF ECG RECORDINGS

ECG recordings are safe. Some people may develop mild irritation due to the adhesive used to hold the electrodes on. The gel may also require washing your hands and chest after the study. Rarely, there

VA FORM JAN 1990 10-1086



| Subject Name: | | Date: |
|-------------------------|---------------------------------|------------------|
| Subject Initials: | | |
| Principal Investigator: | THOMAS F. NEWTON | VAMC: |
| H-30334 - CARISBAMATE | AS A POTENTIAL TREATMENT FOR AL | COHOL DEPENDENCE |

may be an allergic reaction to ECG

electrode adhesive, which might result in redness or swelling.

## OTHER RISKS AND DISCOMFORTS

During the entry visit you will be asked questions about your medical history and your lifestyle, alcohol and drug use. Some of these questions may be personal, and you may feel uncomfortable or embarrassed. The questions will be asked in a private room such that no one besides the study staff will know your answers.

Visits to the study center for study procedures may be time consuming and inconvenient. Your participation in the study will last about 8 days.

#### Risks associated with privacy

This study involves sensitive and confidential issues regarding drug and alcohol use. Although we will take all precautions necessary to safeguard your privacy, there are risks associated with invasion of privacy and breaches of confidentiality. Examples are embarrassment within ones professional or social group (stigmatization), loss of employability and insurability, or criminal prosecution, and disruption of family relationships.

You should be aware that insurance companies and employers may be interested in knowing if you have ever participated in a research study. In the course of applying for certain types of insurance (e.g., medical, life insurance, or disability insurance), you may be asked to sign release forms that authorize insurance companies to obtain your medical records from MEDVAMC. We will keep research records containing confidential information about your participation separate from your medical records so that they will be inaccessible to insurance companies who access patient medical records.

### PRIVACY AND CONFIDENTIALITY

The only people who will know that you are a research subject are members of the research team and, if appropriate, your physicians and nurses. To reduce the chance that someone will find out about you staying at the VA, you may use an assumed name in interacting with the research staff; however, your medical record will still reflect your real name. No information about you, or provided by you during the research, will be disclosed to others without your written permission, except if necessary to protect your rights and welfare (for example, if you are injured and need emergency care.)

To help us protect your privacy, we have obtained a Certificate of Confidentiality from the National Institutes of Health. With this Certificate, the researchers cannot be forced to disclose information that may identify you, even by a court subpoena, in any federal, state, or local civil, criminal, administrative, legislative, or other proceedings. The researchers will use the Certificate to resist any demands for information that would identify you, except as explained below.

VA FORM **10-1086** 



| Subject Name: | | Date: |
|---|---|---|
| Subject Initials: | | |
| Principal Investigator: | THOMAS F. NEWTON | VAMC: |
| H-30334 - CARISBAMATI | E AS A POTENTIAL TREATMENT FOR AL | LCOHOL DEPENDENCE |

The Certificate cannot be used to resist a demand for information from personnel of the United States Government that is used for auditing or evaluation of Federally funded projects or for information that must be disclosed in order to meet the requirements of the federal Food and DrugAdministration (FDA). You should understand that a Certificate of Confidentiality does not prevent you or a member of your family from voluntarily releasing information about yourself or your involvement in this research. If an insurer, employer, or other person obtains your written consent to receive research information, then the researchers may not use the Certificate to withhold that information.

The Certificate of Confidentiality does not prevent the researchers from disclosing voluntarily, without your consent, information that would identify you as a participant in the research project under some circumstances, such as communicable diseases or child or elder abuse. The investigator may also report certain communicable diseases to the county board of health, when s/ he first learns that someone has one of the diseases involved. Examples of these diseases include hepatitis B and C, syphilis, and measles.

When the results of the research are published or discussed in conferences, no information will be included that would reveal your identity. Authorized representatives of the Food and DrugAdministration (FDA), and study monitors from the National Institute on DrugAbuse (NIDA) may need to review records of individual subjects. As a result, they may see your name, but they are bound by rules of confidentiality not to reveal your identity to others. The results of this study including laboratory results and clinical information collected during this study will be submitted to the FDA and may be used for research purposes. The results of this study may be published but will not personally identify you. All records will be kept in locked storage locations that will be accessible only to authorized study personnel. Also, because this research is regulated by the Food and DrugAdministration and sponsored NIDA, staff from these and other DHHS agencies may review records that identify you. However, it is the policy of these agencies and this investigator that every attempt will be made to resist demands to release information that identifies you.

There may be unknown risks or discomforts involved. Study staff will update you in a timely way on any new information that may affect your decision to stay in the study.

#### **Potential Benefits**

You will receive no direct benefit from your participation in this study. However, your participation may help the investigators better understand the usefulness of carisbamate for treating alcohol dependence..

#### **Alternatives**

The following alternative procedures or treatments are available if you choose not to participate in this study: Various behavioral treatment programs are available if you choose not to participate in this study, including counseling, residential programs, and twelve step programs.

VA FORM **10-1086** 

| Department of Vete | VA RESEARCH CONS | SENT FORM |
|------------------------|------------------|-----------|
| Subject Name: | | Date: |
| Subject Initials: | | |
| rincipal Investigator: | THOMAS F. NEWTON | VAMC: |

## Investigator Withdrawal of Subject from a Study

The investigator may withdraw you from participating in this research if circumstances arise which warrant doing so. You may have to drop out of the study even if you would like to continue. You will be removed from the study without your

consent for any of the following reasons:

The investigator decides that continuing in the study would be harmful to you.

You secretly use alcohol or illicit drugs while on the study.

You need to take medications that are not allowed while on this study.

You are unable to keep appointments or complete study procedures as instructed.

You have a bad reaction to your study drug such that you can no longer continue to take them.

You no longer meet the eligibility requirements for this study.

The study is canceled by the Food and Drug Administration, or Baylor College of Medicine.

The investigator will make the decision and let you know if it is not possible for you to continue. The decision may be made either to protect your health and safety, or because it is part of the research plan that people who develop certain conditions may not continue to participate.

## **Subject Costs and Payments**

You will not be asked to pay any costs related to this research.

VA FORM JAN 1990 10-1086

| Subject Name: | | Date: |
|---|---|---|
| Subject Initials: | | |
| Principal Investigator: | THOMAS F. NEWTON | VAMC: |
| H-30334 - CARISBAMATE | AS A POTENTIAL TREATMENT FOR ALCOHOL DE | EPENDENCE |

You will be paid \$40 in gift certificates for the completion of the screening. \$50/day is the average compensation provided across the 8 study days. The compensation increases over the course of the study to compensate for the increasing difficulty you may have in abstaining from alcohol use. The payment schedule is shown below. You can earn up to \$440 if you complete the entire study (including the screening payment). You will be paid by check at the time of your discharge.

Phase 1

Day 1 - \$20

Day 2 - \$40

Day 3 - \$60

Day 4 - \$80

total \$200

Phase 2

Day 1 - \$20

Day 2 - \$30

Day 3 - \$40

Day 4 - \$110

total \$200

# **Research Related Injury**

If you are injured as a direct result of research procedures you will receive treatment as necessary at no cost to you.

The MED-VAMC and NIDA do not provide any other form of compensation for injury.

JAN 1990

10-1086

Last Amendment: 8/26/2013 BCM Approval from June 13, 2017 to June 12, 2018



| Subject Name: | | Date: |
|---|---|---|
| Subject Initials: | | |
| Principal Investigator: | THOMAS F. NEWTON | VAMC: |
| H-30334 - CARISBAMAT | E AS A POTENTIAL TREATMENT FOR A | LCOHOL DEPENDENCE |

## **Subject's Rights**

Your signature on this consent form means that you have received the information about this study and that you agree to volunteer for this research study.

You will be given a copy of this signed form to keep. You are not giving up any of your rights by signing this form. Even after you have signed this form, you may change your mind at any time. Please contact the study staff if you decide to stop taking part in this study.

If you choose not to take part in the research or if you decide to stop taking part later, your benefits and services will stay the same as before this study was discussed with you. You will not lose these benefits, services, or rights.

Your Health Information

Your signature on this form means that you give permission for the use and disclosure of your protected health information for this research study. Federal law requires that the Michael E. Debakey Veterans Affairs Medical Center protect health information linked to your identity. The procedures section above provides the specific information and the person(s) who would use or disclose it.

If you decide not to give your permission for the use and disclosure of your protected health information as we have described for this study, you will receive access to the same treatment, payment, enrollment or eligibility for benefits as you normally would.

People who give medical care and ensure quality from the institutions where the research is being done, the sponsor(s) listed in the sections above, representatives of the sponsor, agents of the Food and Drug Administration, and regulatory agencies such as the U.S. Department of Health and Human Services will be allowed to look at sections of your medical and research records related to this study. Because of the need for the investigator and study staff to release information to these parties, complete privacy cannot be guaranteed. There may be a risk of loss of confidentiality by participating in this study.

If you decide to take part in the study, your protected health information will not be given out except as allowed by the regulations or as described in this form. The results of the data from the study may be published. However, you will not be identified by name. People who receive your protected health information may not be required by Federal privacy laws to protect it and may share your information with others without your permission, if permitted by laws governing them.

You may decide that you no longer allow protected health information that identifies you to be used or disclosed for this research study. Contact the study staff to tell them of this decision, and they will give

VA FORM JAN 1990 10-1086



| Subject Name: | | Date: |
|---|---|---|
| Subject Initials: | | |
| Principal Investigator: | THOMAS F. NEWTON | VAMC: |
| H-30334 - CARISBAMAT | E AS A POTENTIAL TREATMENT FOR ALCOH | IOI DEPENDENCE |

you an address so that you can inform the investigator in writing. The investigator will honor this decision unless the researchers have already acted in reliance on your information. Then it will not be possible to honor your decision in this way.

The people listed above will be able to access your information for as long as they need to, even after the study is completed.

The investigator, THOMAS F. NEWTON, and/or someone he/she appoints in his/her place will try to answer all of your questions. If you have questions or concerns at any time, or if you need to report an injury related to the research, you may speak with a member of the study staff: THOMAS F. NEWTON at 713-791-1414 x6498 during the day, Richard De La Garza, Ph.D. at 713-791-1414 x6020 during the day. After hours you can reach the study team at 877-228-5777. If you have any questions about the study or wish to inquire regarding your eligibility status, please call us at 877-228-5777. This is our 24 hour study hotline number. A staff member will be able to answer any questions you may have

Members of the Institutional Review Board for Baylor College of Medicine and Affiliated Hospitals (IRB) can also answer your questions and concerns about your rights as a research subject. The IRB office number is (713) 798-6970. Call the IRB office if you would like to speak to a person independent of the investigator and research staff for complaints about the research, if you cannot reach the research staff, or if you wish to talk to someone other than the research staff.

Under Federal Regulations, the VA Medical facility shall provide necessary medical treatment to you as a research subject injured as a result by participation in a research project approved by a VA Research and Development Committee and conducted under the supervision of one or more VA employees. This requirement does not apply to treatment for injuries that result from non-compliance by a research subject with study procedures. If you sustain an injury as a direct result of your study participation, medical care will be provided by the Michael E. DeBakey VA Medical Center. The Department of Veterans Affairs does not normally provide any other form of compensation for injury. You do not waive any liability rights for personal injury by signing this form.

You may withdraw from this study at any time without penalty or loss of VA or other benefits to which you are entitled. Your participation will not affect the way you now pay for medical care at the VAMC. If you would like to verify the validity of the study and authorized contacts, you may speak with the Michael E. DeBakey Veterans Affairs Medical Center Research Office at 713-794-7918 or 713-794-7566.

VA FORM **10-1086** 

| Subject Name: | | Date: |
|---|---|---|
| Subject Initials: | | |
| Principal Investigator: | THOMAS F. NEWTON | VAMC: |
| | E AS A POTENTIAL TREATMENT FO | |
| Signing this consent form that your questions have I | indicates that you have read this conceen answered to your satisfaction, an study. You will receive a copy of thi | sent form (or have had it read to you nd that you voluntarily agree to |

Date

VA FORM JAN 1990 **10-1086** 

Last Amendment: 8/26/2013

Witness